CLINICAL TRIAL: NCT00591578
Title: A Double-Blind, Randomized, Parallel-Group Study to Compare the Efficacy and Safety of TAK-491 With Valsartan in Subjects With Essential Hypertension
Brief Title: Efficacy and Safety Comparison of Azilsartan Medoxomil to Valsartan in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-491_301; U1111-1113-9238 (Registry Identifier: WHO)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: Blood pressure; blood pressure monitoring, ambulatory
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil; azilsartan; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil
- Azilsartan Medoxomil 80 mg QD (Experimental)
  Interventions: Drug: Azilsartan Medoxomil
- Valsartan 320 mg QD (Active Comparator)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Azilsartan Medoxomil — Azilsartan Medoxomil 20 mg, tablets, orally, once daily for 2 weeks; titrated to 40 mg, tablets, orally, once daily for up to 22 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 40 mg QD
Drug: Azilsartan Medoxomil — Azilsartan Medoxomil 20 mg, tablets, orally, once daily for 2 weeks; titrated to 80 mg, tablets, orally, once daily for up to 22 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 80 mg QD
Drug: Valsartan — Valsartan 80 mg, tablets, orally, once daily for 2 weeks; titrated to 320 mg, tablets, orally, once daily for up to 22 weeks.
  Other Names: Diovan
  Arms: Valsartan 320 mg QD

SUMMARY:
The purpose of this study is to compare the efficacy and safety of TAK-491 (azilsartan medoxomil), once daily (QD), to valsartan in participants with essential hypertension.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. According to the World Health Organization (WHO), hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of antihypertensive treatments, hypertension remains inadequately controlled; only about one-third of patients continue to maintain control successfully.

This study is being conducted to determine whether administration of azilsartan medoxomil in subjects with essential hypertension is more efficacious in reducing systolic blood pressure than valsartan.

Study participation is anticipated to be approximately 7 months. Outside of the study center, participants will be required to wear an ambulatory blood pressure monitoring device at 24 hour intervals.

Following completion of the 6-month double-blind treatment period, all available subjects will be offered the option to continue in a 28-week extension study with open-label azilsartan medoxomil 40 mg.

For the extension study, participants will take azilsartan medoxomil 40 mg, tablets, orally, once daily for up to 28 weeks. Hydrochlorothiazide 12.5 mg or 25 mg or any other antihypertensive (except angiotensin II receptor blockers) may be added in a step-wise fashion to maintain blood pressure within target <140/90 mmHg for non-diabetic subjects and <130/80 mmHg for diabetic subjects

ELIGIBILITY:
Inclusion Criteria

1. Essential hypertension (defined as sitting trough clinic systolic blood pressure between 150 and 180 mm Hg inclusive at Day minus 1 and 24-hour mean systolic blood pressure between 130 and 170 mm Hg inclusive at Day 1).
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
3. Clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory or the results are deemed not clinically significant for inclusion into this study by the investigator.
4. Willing to discontinue current antihypertensive medications at the Screening Day minus 21 visit. If the subject is on amlodipine prior to Screening, the subject is willing to discontinue this medication at Screening Day minus 28.

Exclusion Criteria

1. Sitting trough clinic diastolic blood pressure greater than 114 mm Hg at Day minus 1.
2. The subject has a baseline 24-hour ambulatory blood pressure monitor reading of insufficient quality.
3. Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication.
4. Hypersensitive to angiotensin II receptor blockers.
5. Recent history (within the last 6 months) of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
6. Clinically significant cardiac conduction defects (eg, 3rd degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation or flutter).
7. Hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
8. Secondary hypertension of any etiology.
9. Non-compliant (less than 70% or greater than 130%) with study medication during placebo run-in period.
10. Severe renal dysfunction or disease (based on calculated creatinine clearance less than 30 mL per min/1.73m2) at Screening.
11. Known or suspected unilateral or bilateral renal artery stenosis.
12. History of drug or alcohol abuse within the past 2 years.
13. Previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin).
14. Type 1 or poorly controlled type 2 diabetes mellitus (glycosylated hemoglobin greater than 8.0%) at Screening.
15. Hyperkalemia as defined by the central laboratory normal reference range at Screening.
16. Upper arm circumference less than 24 cm or greater than 42 cm.
17. Works night (3rd) shift (defined as 11PM to 7AM).
18. Alanine aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice at Screening.
19. Currently is participating in another investigational study or has participated in an investigational study within 30 days prior to randomization.
20. Any other serious disease or condition at Screening (or Randomization) that would compromise subject safety, might affect life expectancy, or make it difficult to successfully manage and follow the subject according to the protocol.
21. Randomized in a previous azilsartan medoxomil study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director Clinical Science, Study Director — Takeda
Locations (88):
- United States (77):
  - Huntsville, Alabama
  - Glendale, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tuscon, Arizona
  - Beverly Hills, California
  - Burbank, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Paramount, California
  - San Diego, California
  - Santa Monica, California
  - Spring Valley, California
  - Tustin, California
  - Vista, California
  - Westlake Village, California
  - Ridgefield, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Morton, Illinois
  - Park Ridge, Illinois
  - Avon, Indiana
  - Bloomington, Indiana
  - Crestview Hills, Kentucky
  - Baltimore, Maryland
  - Columbia, Maryland
  - Brockton, Massachusetts
  - West Yarmouth, Massachusetts
  - Ann Arbor, Michigan
  - City of Saint Peters, Missouri
  - Florissant, Missouri
  - Kansas City, Missouri
  - Washington, Missouri
  - Wentzville, Missouri
  - Charlotte, North Carolina
  - Salisbury, North Carolina
  - Shelby, North Carolina
  - Cincinnati, Ohio
  - Delaware, Ohio
  - Mogadore, Ohio
  - Willoughby Hills, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Bridgeville, Pennsylvania
  - Downingtown, Pennsylvania
  - Jenkintown, Pennsylvania
  - Lansdale, Pennsylvania
  - Charleston, South Carolina
  - Spartanburg, South Carolina
  - Kingsport, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Pearland, Texas
  - Rosenberg, Texas
  - San Antonio, Texas
  - Riverton, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Arlington, Virginia
  - Burke, Virginia
  - Norfolk, Virginia
  - Lakewood, Washington
  - Port Richard, Washington
  - Menomonee Falls, Wisconsin
- Chile (2):
  - Santiago
  - Temuco
- Mexico (7):
  - Cabo San Lucas
  - Colonia Escandón
  - Culiacán
  - Mexico City
  - Monterrey Nuevo Leon
  - Morelia
  - Querétaro
- Peru (2):
  - Chiclayo
  - Lima

REFERENCES:
- [Result] Sica D, White WB, Weber MA, Bakris GL, Perez A, Cao C, Handley A, Kupfer S. Comparison of the novel angiotensin II receptor blocker azilsartan medoxomil vs valsartan by ambulatory blood pressure monitoring. J Clin Hypertens (Greenwich). 2011 Jul;13(7):467-72. doi: 10.1111/j.1751-7176.2011.00482.x. Epub 2011 Jun 20. PMID 21762358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 103 investigative sites from 09 November 2007 to 03 September 2009 (double-blind phase) and 04 March 2009 to 13 March 2010 (open-label extension phase). A total of 984 participants were randomized into the double-blind treatment phase, of which 170 participants entered into the open-label extension phase.
Pre-assignment Details: Participants with essential hypertension were enrolled in one of three, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for 2 weeks; titrated to 40 mg, tablets, orally, once daily for up to 22 weeks.
  Open Label Extension: At Week 24/completion of the double-blind treatment phase, participants could elect to continue in 28 week, open-label extension (OLE) phase. All participants who elected to participate in the OLE phase initiated treatment with azilsartan medoxomil 40 mg, tablets, orally, independent of their double-blind treatment assignment. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for 2 weeks; titrated to 80 mg, tablets, orally, once daily for up to 22 weeks.
  Open Label Extension: At Week 24/completion of the double-blind treatment phase, participants could elect to continue in 28 week, open-label extension (OLE) phase. All participants who elected to participate in the OLE phase initiated treatment with azilsartan medoxomil 40 mg, tablets, orally, independent of their double-blind treatment assignment. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
- Valsartan 320 mg QD: Valsartan 80 mg, tablets, orally, once daily for 2 weeks; titrated to 320 mg, tablets, orally, once daily for up to 22 weeks.
  Open Label Extension: At Week 24/completion of the double-blind treatment phase, participants could elect to continue in 28 week, open-label extension (OLE) phase. All participants who elected to participate in the OLE phase initiated treatment with azilsartan medoxomil 40 mg, tablets, orally, independent of their double-blind treatment assignment. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
Period: Double-Blind Treatment Phase
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Started | 327 | 329 | 328 (Two participants randomized but not treated.)
Completed | 249 | 249 | 244
Not Completed | 78 | 80 | 84
Not completed — Adverse Event | 20 | 26 | 19
Not completed — Protocol Violation | 3 | 2 | 3
Not completed — Lost to Follow-up | 12 | 12 | 11
Not completed — Withdrawal by Subject | 22 | 22 | 22
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Lack of Efficacy | 16 | 9 | 25
Not completed — Other | 4 | 9 | 4
Period: Open-Label Extension Phase
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Started | 55 | 115 | 0
Completed | 49 | 105 | 0
Not Completed | 6 | 10 | 0
Not completed — Adverse Event | 3 | 5 | 0
Not completed — Lost to Follow-up | 1 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for 2 weeks; titrated to 40 mg, tablets, orally, once daily for up to 22 weeks.
  Open Label Extension: Azilsartan medoxomil 40 mg, tablets, orally, once daily for 28 weeks. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
  Open Label Extension: Azilsartan medoxomil 40 mg, tablets, orally, once daily for 28 weeks. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for 2 weeks; titrated to 80 mg, tablets, orally, once daily for up to 22 weeks.
  Open Label Extension: Azilsartan medoxomil 40 mg, tablets, orally, once daily for 28 weeks. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
  Open Label Extension: Azilsartan medoxomil 40 mg, tablets, orally, once daily for 28 weeks. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
- Valsartan 320 mg QD: Valsartan 80 mg, tablets, orally, once daily for 2 weeks; titrated to 320 mg, tablets, orally, once daily for up to 22 weeks.
  Open Label Extension: Azilsartan medoxomil 40 mg, tablets, orally, once daily for 28 weeks. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Total
Number analyzed (Participants) | 327 | 329 | 328 | 984
Age, Customized [Number; unit: participants]
  <45 years (Double Blind Phase) | 43 | 39 | 31 | 113
  Between 45 and 64 years (Double Blind Phase) | 181 | 208 | 199 | 588
  ≥65 years (Double Blind Phase) | 103 | 82 | 98 | 283
  <45 years (Open Label Phase) | 10 | 8 | 0 | 18
  Between 45 and 64 years (Open Label Phase) | 25 | 68 | 0 | 93
  ≥65 years (Open Label Phase) | 20 | 39 | 0 | 59
Sex/Gender, Customized [Number; unit: participants]
  Female (Double Blind Phase) | 163 | 160 | 152 | 475
  Male (Double Blind Phase) | 164 | 169 | 176 | 509
  Female (Open Label Phase) | 34 | 57 | 0 | 91
  Male (Open Label Phase) | 21 | 58 | 0 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for 2 weeks; titrated to 40 mg, tablets, orally, once daily for up to 22 weeks.
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for 2 weeks; titrated to 80 mg, tablets, orally, once daily for up to 22 weeks.
- Valsartan 320 mg QD: Valsartan 80 mg, tablets, orally, once daily for 2 weeks; titrated to 320 mg, tablets, orally, once daily for up to 22 weeks.
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -14.93 (0.698) | -15.32 (0.715) | -11.29 (0.707)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value presented. Overall 0.05 level of significance for multiple comparisons controlled using stepwise testing procedure; Mean Difference (Final Values) = -3.64, 95% CI 2-sided [-5.59 to -1.69]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Unadjusted p-value presented. Overall 0.05 level of significance for multiple comparisons controlled using stepwise testing procedure; Mean Difference (Final Values) = -4.03, 95% CI 2-sided [-6.01 to -2.06]

2. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Systolic Blood Pressure.
Description: The change in mean trough clinic sitting systolic blood pressure measured at final visit or week 24 relative to baseline. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 323 | 311 | 322
mmHg | -14.86 (0.948) | -16.92 (0.966) | -11.59 (0.949)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.015, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). The unadjusted p-value is presented; Mean Difference (Final Values) = -3.27, 95% CI 2-sided [-5.90 to -0.63]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.34, 95% CI 2-sided [-8.00 to -2.68]

3. Secondary Outcome: Change From Baseline in the 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -9.23 (0.459) | -9.77 (0.470) | -7.07 (0.465)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-3.44 to -0.88]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.69, 95% CI 2-sided [-3.99 to -1.40]

4. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Diastolic Blood Pressure
Description: The change in mean trough clinic sitting diastolic blood pressure measured at final visit or week 24 relative to baseline. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 323 | 311 | 322
mmHg | -7.16 (0.554) | -7.41 (0.565) | -4.65 (0.555)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.52, 95% CI 2-sided [-4.06 to -0.98]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.76, 95% CI 2-sided [-4.32 to -1.21]

5. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -15.39 (0.732) | -15.80 (0.749) | -11.91 (0.741)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.49, 95% CI 2-sided [-5.53 to -1.44]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.90, 95% CI 2-sided [-5.96 to -1.83]

6. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: as for outcome 5
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -9.61 (0.493) | -10.11 (0.504) | -7.44 (0.499)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.17, 95% CI 2-sided [-3.54 to -0.79]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.67, 95% CI 2-sided [-4.06 to -1.28]

7. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -13.31 (0.777) | -13.95 (0.795) | -9.52 (0.786)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.79, 95% CI 2-sided [-5.96 to -1.62]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.44, 95% CI 2-sided [-6.63 to -2.24]

8. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -8.06 (0.526) | -8.90 (0.539) | -6.06 (0.533)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.00, 95% CI 2-sided [-3.48 to -0.53]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.84, 95% CI 2-sided [-4.33 to -1.35]

9. Secondary Outcome: Change From Baseline in the 12-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -15.64 (0.764) | -16.20 (0.782) | -12.20 (0.774)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.44, 95% CI 2-sided [-5.57 to -1.30]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.01, 95% CI 2-sided [-6.16 to -1.85]

10. Secondary Outcome: Change From Baseline in the 12-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean diastolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -9.70 (0.522) | -10.26 (0.534) | -7.53 (0.528)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.18, 95% CI 2-sided [-3.63 to -0.72]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-4.20 to -1.25]

11. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -13.74 (0.851) | -13.83 (0.871) | -10.36 (0.861)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.38, 95% CI 2-sided [-5.76 to -1.00]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.47, 95% CI 2-sided [-5.87 to -1.06]

12. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean diastolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 284 | 271 | 277
mmHg | -9.37 (0.617) | -9.65 (0.632) | -7.06 (0.625)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.009, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.31, 95% CI 2-sided [-4.04 to -0.59]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.59, 95% CI 2-sided [-4.34 to -0.84]

13. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Systolic Blood Pressure Response, Defined as < 140 mm Hg and/or Reduction From Baseline ≥ 20 mm Hg.
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at week 24, defined as less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 323 | 311 | 322
percentage of participants | 56.0 | 59.2 | 46.9
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.016, Regression, Logistic — P-value for response criteria for systolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Includes only those participants with a baseline and at least one post-baseline value; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.07 to 2.00]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Includes only those participants with a baseline and at least one post-baseline value; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.19 to 2.23]

14. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic Blood Pressure Response, Defined as < 90 mm Hg and/or Reduction From Baseline ≥ 10 mm Hg.
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at week 24, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 323 | 311 | 322
percentage of participants | 72.4 | 74.0 | 65.8
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.041, Regression, Logistic — P-value for response criteria for diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic diastolic blood pressure as a covariate. The unadjusted p-value is presented; Includes only those participants with a baseline and at least one post-baseline value; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.02 to 2.10]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.015, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Includes only those participants with a baseline and at least one post-baseline value; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.09 to 2.28]

15. Secondary Outcome: Percentage of Participants Who Achieve Both a Clinic Diastolic and Systolic Blood Pressure Response.
Description: Percentage of participants who achieve both a clinic diastolic and systolic blood pressure response measured at week 24, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg AND less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Diastolic and systolic blood pressure is based on the arithmetic mean of the 3 sitting blood pressure measurements.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD
Number analyzed (Participants) | 323 | 311 | 322
percentage of participants | 50.2 | 54.7 | 41.3
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.018, Regression, Logistic — P-value for joint response criteria for systolic blood pressure and diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Includes only those participants with a baseline and at least one post-baseline value; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.07 to 1.99]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Includes only those participants with a baseline and at least one post-baseline value; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.24 to 2.33]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Open Label Extension: Azilsartan medoxomil 40 mg, tablets, orally, independent of participant's double-blind treatment assignment. Investigators may have added, in a step-wise fashion, hydrochlorothiazide 12.5 mg, followed by hydrochlorothiazide 25 mg, followed by other antihypertensive medications (except angiotensin II receptor blockers) as needed to achieve target blood pressure (<140/90 mm Hg or <130/80 mm Hg for diabetics).
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Open Label Extension
Serious Adverse Events (participants affected / at risk) | 8/327 | 5/329 | 8/326 | 4/170
Other Adverse Events (participants affected / at risk) | 77/327 | 74/329 | 53/326 | 16/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD (N=327) | Azilsartan Medoxomil 80 mg QD (N=329) | Valsartan 320 mg QD (N=326) | Open Label Extension (N=170)
Silent myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD (N=327) | Azilsartan Medoxomil 80 mg QD (N=329) | Valsartan 320 mg QD (N=326) | Open Label Extension (N=170)
Urinary tract infection (Infections and infestations) | 26 | 25 | 16 | 10
Dizziness (Nervous system disorders) | 27 | 29 | 15 | 8
Headache (Nervous system disorders) | 33 | 29 | 28 | 9

LIMITATIONS AND CAVEATS:
For the Non-Serious Adverse Event Table, the total number of participants affected is based on the AEs with ≥5% in each phase, calculated separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.